CLINICAL TRIAL: NCT07074327
Title: Phase 1, Open-label Study to Evaluate the Effect of VX-407 on the Pharmacokinetics of Oral Contraceptives in Healthy Subjects
Brief Title: Effects of VX-407 on the Pharmacokinetics of Oral Contraceptives in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VX24-407-006
Record Dates: First submitted 2025-07-09; First posted 2025-07-20 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Keywords: Oral contraceptives; Drug interaction; Pharmacokinetics
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: VX-407 With Levonorgestrel/Ethinyl Estradiol (LNG/EE) (Experimental): Participants will receive a single dose of LNG/EE on Days 1 and 21 in fasted state. Participants will also receive VX-407 every 12 hours (q12h) from Days 8 through 26 in fasted state.
  Interventions: Drug: VX-407; Drug: LNG/EE
- Part B (Optional): VX-407 With Norgestimate/Ethinyl Estradiol (NGM/EE) (Experimental): Participants will receive a single dose of NGM/EE on Days 1 and 23 in fasted state. Participants will also receive VX-407 q12h from Days 10 through 30 in fasted state.
  Interventions: Drug: VX-407; Drug: NGM/EE
- Part C (Optional): VX-407 With Norethindrone/Ethinyl Estradiol (NET/EE) (Experimental): Participants will receive a single dose of NET/EE on Days 1 and 19 in fasted state. Participants will also receive VX-407 q12h from Days 6 through 22 in fasted state.
  Interventions: Drug: VX-407; Drug: NET/EE
- Part D (Optional): VX-407 With Drospirenone/Ethinyl Estradiol (DRSP/EE) (Experimental): Participants will receive a single dose of DRSP/EE on Days 1 and 21 in fasted state. Participants will also receive VX-407 q12h from Days 8 through 26 in fasted state.
  Interventions: Drug: VX-407; Drug: DRSP/EE

INTERVENTIONS:
Drug: VX-407 — Suspension for oral administration.
Drug: LNG/EE — Combination Tablets for Oral Administration.
  Arms: Part A: VX-407 With Levonorgestrel/Ethinyl Estradiol (LNG/EE)
Drug: NGM/EE — Combination Tablets for Oral Administration.
  Arms: Part B (Optional): VX-407 With Norgestimate/Ethinyl Estradiol (NGM/EE)
Drug: NET/EE — Combination Tablets for Oral Administration.
  Arms: Part C (Optional): VX-407 With Norethindrone/Ethinyl Estradiol (NET/EE)
Drug: DRSP/EE — Combination Tablets for Oral Administration.
  Arms: Part D (Optional): VX-407 With Drospirenone/Ethinyl Estradiol (DRSP/EE)

SUMMARY:
The purpose of the study is to evaluate the effect of VX-407 on the pharmacokinetics of levonorgestrel (LNG) and ethinyl estradiol (EE), norgestimate (NGM) and EE, norethindrone (NET) and EE and drospirenone (DRSP) and EE. Also, to evaluate the safety and tolerability of co-administration of VX-407 with LNG/EE, NGM/EE, NET/EE and DRSP/EE.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 30.0 kilogram per meter square (kg/m^2)
* A total body weight of greater than (>) 50 kg
* Nonsmoker or ex-smoker for at least 12 months before screening
* Oral contraceptive naïve or able to comply with 28-day or 5 half-lives (whichever is greater) washout before the start of Period 1 (6-month washout for Depo-Provera)

Exclusion Criteria:

* History of febrile illness within 5 days before the first dose of study drug
* Relative contraindications to hormonal estrogen therapy that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant
* Any condition possibly affecting drug absorption, distribution, metabolism, or excretion
* Pregnant, nursing, or planning to become pregnant during the study or within 90 days after the last dose of study drug
* Menopausal, post-menopausal, or documented bilateral oophorectomy and/or hysterectomy
* Previously received study drug in this study

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-06-29 (Estimated); Study Completion 2026-07-04 (Estimated)

PRIMARY OUTCOMES:
Part A: Maximum Observed Plasma Concentration (Cmax) of LNG and EE in the Absence and Presence of VX-407 | From Day 1 up to Day 7 and Day 21 up to Day 27
Part A: Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of LNG and EE in the Absence and Presence of VX-407 | From Day 1 up to Day 7 and Day 21 up to Day 27
Part B (Optional): Cmax of Norelgestromin (NGMN) and Norgestrel (NG) (Active Metabolites of NGM) and EE in the Absence and Presence of VX-407 | From Day 1 up to Day 9 and Day 23 up to Day 31
Part B (Optional): AUC0-inf of NGMN and NG (Active Metabolites of NGM) and EE in the Absence and Presence of VX-407 | From Day 1 up to Day 9 and Day 23 up to Day 31
Part C (Optional): Cmax of NET and EE in the Absence and Presence of VX-407 | From Day 1 up to Day 5 and Day 19 up to Day 23
Part C (Optional): AUC0-inf of NET and EE in the Absence and Presence of VX-407 | From Day 1 up to Day 5 and Day 19 up to Day 23
Part D (Optional): Cmax of DRSP and EE in the Absence and Presence of VX-407 | From Day 1 up to Day 7 and Day 21 up to Day 27
Part D (Optional): AUC0-inf of DRSP and EE in the Absence and Presence of VX-407 | From Day 1 up to Day 7 and Day 21 up to Day 27

SECONDARY OUTCOMES:
Part A: Safety and Tolerability as Assessed by Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 36
Part B (Optional): Safety and Tolerability as Assessed by Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 40
Part C (Optional): Safety and Tolerability as Assessed by Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 32
Part D (Optional): Safety and Tolerability as Assessed by Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 36
Part A: Cmax of VX-407 | Days 9, 15 and 21 up to Day 27
Part A: AUC0-inf of VX-407 | Days 9, 15 and 21 up to Day 27
Part B (Optional): Cmax of VX-407 | Days 11, 17 and 23 up to Day 31
Part B (Optional): AUC0-inf of VX-407 | Days 11, 17 and 23 up to Day 31
Part C (Optional): Cmax of VX-407 | Days 7, 13 and 19 up to Day 23
Part C (Optional): AUC0-inf of VX-407 | Days 7, 13 and 19 up to Day 23
Part D (Optional): Cmax of VX-407 | Days 9, 15 and 21 up to Day 27
Part D (Optional): AUC0-inf of VX-407 | Days 9, 15 and 21 up to Day 27

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences - Kansas City, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing